CLINICAL TRIAL: NCT00541372
Title: The Influence of the Needle Length on Long Term Glycaemic Control in Insulin Using Obese Diabetic Subjects
Brief Title: Needle Length In Obese Insulin-Using Diabetic Subjects
Acronym: INOBESE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Martini Hospital Groningen (Other)
Responsible Party: B.H.R. Wolffenbuttel, Univ Med Ctr Groningen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BWO-07001
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Needle 5 mm
  Interventions: Device: insulin injection needle size
- 2 (Active Comparator): Needle length 8 mm
  Interventions: Device: insulin injection needle size

INTERVENTIONS:
Device: insulin injection needle size — The intervention in this study is a specific needle with a length of 5 mm and 8 mm to be used with an insulin pen.

SUMMARY:
For the administration of insulin, different needles are available with a length from 5 to 12.7mm. Insulin injections with a needle of 8 mm is injected in a lifted skinfold, a 5 mm needle can by used without lifting a skinfold (1). In the Netherlands obese people (BMI ≥ 30) are usually advised to use an 8mm or even longer needle (1). Increased BMI and the thickness of the subcutaneous tissue slow insulin absorption (2, 3, 4), possibly related to reduced subcutaneous blood flow. Furthermore, the capillaries are located just under the skin and between the fat and muscle layer. This could possibly determine the absorbing speed (2). It is not know if the administration of insulin with a 5mm needle by obese people has a different influence on the HbA1c compared to longer needles. The hypothesis of this study is that for the purpose of insulin injections, a 5 mm needle can be used without negative effects on metabolic parameters in patients with Diabetes Mellitus (DM) and a Body Mass Index (BMI) ≥ 30.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients diagnosed with type 1 and type 2 diabetes mellitus, treated with insulin injections for at least one year and:

  * using an insulin pen
  * a BMI > 30 kg/m2
  * a skinfold thickness of >10 mm at the injection sites
  * stable glycaemic control, with HbA1c between 6 and 10%
  * capable of reading the written information
  * prepared to, and capable of signing an informed consent

Exclusion Criteria:

* Patients who:

  * change their own insulin dosage and are not prepared to keep a record of these changes
  * have hypoglycaemia unawareness
  * are pregnant or wish to become pregnant
  * have a BMI < 30 kg/m2
  * have a skinfold thickness <10mm
  * have skin problems including lipodystrophy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Preference of the patient and amount of experienced hypoglycaemic events, bruises, backflow of insulin, bleeding and pain (VAS-scale) | 4 months

SECONDARY OUTCOMES:
HbA1c levels 1,5 anhydroglucitol and fructosamine levels Insulin dose | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce HR Wolffenbuttel, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Kreugel G, Keers JC, Kerstens MN, Wolffenbuttel BH. Randomized trial on the influence of the length of two insulin pen needles on glycemic control and patient preference in obese patients with diabetes. Diabetes Technol Ther. 2011 Jul;13(7):737-41. doi: 10.1089/dia.2011.0010. Epub 2011 Apr 10. PMID 21476936